CLINICAL TRIAL: NCT06949930
Title: OPTIMIZING ROUTINE DELIVERY OF ESSENTIAL CHILD HEALTH AND NUTRITION PACKAGE THROUGH PRIMARY HEALTH CARE CONTACTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition International (Other)
Collaborators: Kenya Ministry of Health (Other Government); Cheikh Anta Diop University, Senegal (Other); Senegal Ministry of Health (Unknown); Henike Consultants (Unknown)
Responsible Party: Principal Investigator, Daniel Lopez de Romana, Director Research, Innovation, and Evaluation, Nutrition International
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nutrition International
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Coverage of Vitamin A Supplementation; Coverage of Immunization; Feasibility and Fidelity of Implementation
Keywords: VAS; immunization; coverage; hybrid effectiveness-implementation research study; essential child health and nutrition services
MeSH Terms: interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Implementation model aims to optimize health workforce training and supervision, service delivery, health data and information, and leadership and governance as so to maximize VAS coverage and in doing so also improve coverage of other services
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm receives the optimized package of child essential health and nutrition services
  Interventions: Other: Optimized package of child essential health and nutrition services
- Control (Other): The control arm receives the current standard package of health and nutrition services
  Interventions: Other: Standard package of essential child and nutrition services

INTERVENTIONS:
Other: Optimized package of child essential health and nutrition services — Optimized package of child essential health and nutrition services
  Arms: Intervention
Other: Standard package of essential child and nutrition services — Standard package of essential child and nutrition services
  Arms: Control

SUMMARY:
The primary objective of the study is to assess whether optimization of an essential package of health and nutrition services for children under five years of age using vitamin A supplementation touch points (i.e., the implementation model) in selected areas in Kenya and Senegal will increase the coverage of vitamin A supplementation and the coverage of other child health and nutrition services. In addition, the study will also assess the feasibility of the implementation model and the drivers of coverage outcomes.

DETAILED DESCRIPTION:
Background: Countries have made significant progress over the last 20 years in improving child survival with under five mortality rates. Despite this progress, many countries still experience inequalities in the coverage of several essential child health and nutrition services, including vitamin A supplementation (VAS), growth monitoring and promotion (GMP), immunization, and regular nutrition screening for early detection of malnutrition. Optimizing the delivery of an Essential Child Health and Nutrition Package ("essential package") may address this issue.

Objective: The primary objective of the study is to assess the effect of optimizing the health system for the delivery of the essential package (the "implementation model"), on the coverage of VAS and on the coverage of immunization (as measured by vaccination for measles). In addition, the study will also assess the feasibility of the implementation model and the drivers of coverage outcomes.

Methods: Target population will be children 12-59 months of age and their caregivers in Kisii County in Kenya and Fatick Region in Senegal. The study will use an effectiveness-research implementation hybrid design with two arms: 1) health system will be optimized to deliver VAS to all children 12-59 months of age using all the routine primary health care (PHC) contact points plus current standard of care (Intervention) and 2) current standard of care (Control). The study will be conducted for a period of 18 months. The optimization model will be implemented for 12 months. Baseline and endline surveys that will collect quantitative and qualitative data will be conducted to assess the coverage of essential child health and nutrition services in both arms from study participants per arm in both baseline and endline surveys and to assess implementation feasibility. Implementation fidelity will be assessed through monthly visits by the research team to health facilities.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children 12-59 months of age
* Health service providers

Exclusion Criteria:

- None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1928 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Children who received their age-appropriate VAS | From enrollment to the end of intervention at 12 months
  The proportion of children 12-59 months of age who received their age-appropriate VAS
Children who are immunized with measles vaccine | From enrollment to the end of intervention at 12 months
  Proportion of children 12-23 months of age who are immunized with one dose of measles (MR1) in Kenya Proportion of children 24-35 months of age who are immunized with the second dose of measles (MR2) in Senegal
Implementation feasibility of new model perceived by health service providers, as assessed by key informant interviews and focus groups | From enrollment to the end of intervention at 12 months
  Feasibility of implementation of the new model as perceived by health service providers will be assessed via key informant interviews and focus groups to enquire on:
  i. Implementation barriers and facilitators ii. Practicality of implementing the optimization model within context and resource availability iii. Program disruption due to the implementation of the model iv. Need for infrastructure to implement the model v. Sustainability of the optimized model.
  All qualitative information will be triangulated to assess feasibility of implementation of the new model
Fidelity of implementing the new model | From enrollment to the end of intervention at 12 months
  Fidelity of implementation will be assessed by measuring:
  i. The proportion of health facilities preparing and using integrated microplans.
  ii. The proportion of supportive supervision visits carried out in an integrated way.
  iii. The proportion of service delivery points providing services in an integrated way
  Fidelity will be achieved if the three parameters score at least 80%.

SECONDARY OUTCOMES:
Co-coverage of VAS and measles vaccine | From enrollment to the end of intervention at 12 months
  Proportion of children 12-23 months of age who have received both their age-appropriate VAS and their age-appropriate vaccines (as measured by measles one) in Kenya Proportion of children 24-35 months of age who have received both their age-appropriate VAS and their age-appropriate vaccines (as measured by measles two) in Senegal
Children screened for malnutrition in the last 6 months | From enrollment to the end of intervention at 12 months
  The proportion of children 12-59 months of age who were screened for malnutrition in the last 6 months
Children who have received growth monitoring service | From enrollment to the end of intervention at 12 months
  The proportion of children 12-59 months who have received growth monitoring service
Children who have received age-appropriate immunizations | From enrollment to the end of intervention at 12 months
  The proportion of children 12-59 months who have received age-appropriate immunizations according to EPI schedule
Caregivers who report receiving more than one service | From enrollment to the end of intervention at 12 months
  The proportion of caregivers of children 12-59 months of age who reported ever receiving more than one of the following services within the Essential Child Health and Nutrition Package during the same visit
Caregivers who indicate are satisfied with the way the services are being delivered | From enrollment to the end of intervention at 12 months
  The proportion of caregivers indicate are satisfied with the way the Essential Child Health and Nutrition Package services are being delivered to their children

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Arabi, M.D., Ph.D., Principal Investigator — Nutrition International; Elijah Mbiti, Ph.D., Principal Investigator — Nutrition International
Locations (2):
- Nutrition International- Kenya, Nairobi, Kenya
- Nutrition International - Senegal, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No